CLINICAL TRIAL: NCT06573060
Title: Impact of Glycemic Variability and Gut Microbiota and Metabolites on the Prognosis of Patients With Type 2 Diabetes Mellitus Combined With Acute Coronary Syndrome
Brief Title: Glycemic Variability, Gut Microbiota, and Prognosis in T2DM With ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: DMACS20240719
Record Dates: First submitted 2024-08-01; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Heart Disease
Keywords: gut microbiome; Type 2 Diabetes mellitus; coronary heart disease; glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faeces and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACS+T2DM: Patients with Type 2 Diabetes Mellitus (T2DM) diagnosed with Acute Coronary Syndrome (ACS) through coronary angiography.
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — Subjects with T2DM and acute coronary syndrome (n=120) were fitted with continuous glucose monitors (CGM) to closely monitor their blood glucose levels continuously for 14 days.

SUMMARY:
Patients with type 2 diabetes mellitus (T2DM) diagnosed with acute coronary syndrome (ACS) by coronary angiography in the Second Affiliated Hospital of Nanchang University were consecutively included in a prospective cohort study. During the acute phase of ACS, blood glucose was monitored using a continuous glucose monitoring system (CGM) for 14 days, and for patients who had been hospitalised for less than 14 days, they continued to wear the CGM for monitoring blood glucose until 14 days after discharge. During this period, stool and serum samples were analysed for multi-omics (16s rRNA sequencing and metabolomics). Subsequently, a follow-up period of at least 1 year was performed to observe the patients for the occurrence of adverse cardiovascular events (MACE) during the follow-up period and to assess the impact of glycaemic variability and gut flora and its metabolites on the prognosis of patients with T2DM combined with ACS.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Type 2 Diabetes Mellitus (T2DM).

Clinical diagnosis of Acute Coronary Syndrome (ACS).

Exclusion Criteria:

History of hemodialysis.

Recent antibiotic use within the past two weeks.

Active malignant tumors.

Pregnancy and breastfeeding.

Inability to wear sensors due to severe skin conditions.

Coagulation disorders, anemia, or abnormal hematocrit levels.

Requirement for MRI during the sensor-wearing period.

Inability to follow study instructions or deemed unsuitable for the trial by the treating clinician/nurse.

Inability to understand informed consent or communicate with researchers due to cognitive decline or mental illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 2023.7-2025.10
  Composite Major Adverse Cardiovascular Events (MACE)

SECONDARY OUTCOMES:
cardiovascular mortality | 2023.7-2025.10
  Deaths due to heart and/or vascular disease. According to the World Health Organisation (WHO) classification, cardiovascular diseases include a wide range of diseases such as coronary heart disease, myocardial infarction, stroke and hypertension.
ACS Recurrence | 2023.7-2025.10
  Refers to the recurrence of a new ACS event after an episode of ACS. Depending on the signs and symptoms, patients can be classified as having STEMI, NSTEMI, or unstable angina.
Angina requiring revascularisation | 2023.7-2025.10
  Presence of indications for coronary revascularisation
Acute decompensated heart failure requiring hospitalisation | 2023.7-2025.10
  Clinical syndrome caused by acute imbalance of oxygen supply and demand due to impaired cardiac function, manifested by dyspnoea, pulmonary oedema and peripheral oedema. The patient's condition is severe enough to require hospitalisation.
Strokes requiring hospitalisation | 2023.7-2025.10
  An acute disease with sudden defects in brain function, such as sudden motor, sensory, speech, and vision disorders. The patient's condition is serious enough to require hospitalisation for treatment and observation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Jiao, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
Privacy and confidentiality issues: Participants' data may contain sensitive personal information. Sharing this data could lead to privacy breaches, violating data protection regulations (such as GDPR).

REFERENCES:
- [Background] Kosiborod M, Rathore SS, Inzucchi SE, Masoudi FA, Wang Y, Havranek EP, Krumholz HM. Admission glucose and mortality in elderly patients hospitalized with acute myocardial infarction: implications for patients with and without recognized diabetes. Circulation. 2005 Jun 14;111(23):3078-86. doi: 10.1161/CIRCULATIONAHA.104.517839. Epub 2005 Jun 6. PMID 15939812
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967